CLINICAL TRIAL: NCT04347031
Title: An Open Randomized Study of the Effectiveness of the Drug Mefloquine, Tablets 250 mg, Produced by FSUE SPC "Farmzashita" of the Federal Medical Biological Agency, FMBA of Russia (Russia) for the Treatment of Patients With COVID19
Brief Title: A Study of the Effectiveness of an Off Label Mefloquine Use for the Treatment of Patients With COVID19
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Burnasyan Federal Medical Biophysical Center (Other Government)
Responsible Party: Principal Investigator, Tatyana Astrelina, MD PhD, DSc (medicine), Head of Center for Biomedical Technologies State Research Center Burnasyan Federal Medical Biophysical Center FMBA of Russia, Burnasyan Federal Medical Biophysical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FL-01/20
Record Dates: First submitted 2020-04-07; First posted 2020-04-15 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Pneumonia, Viral; Respiratory Failure
MeSH Terms: conditions — Pneumonia, Viral; Respiratory Insufficiency | interventions — Mefloquine; Hydroxychloroquine; Azithromycin; tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group 1 cohort 1 (Experimental): 80 patients who receive Mefloquine prescribed according to the following scheme:
  * 1st day: 750 mg of mefloquine per day, inside, in tablets of 250 mg 3 times a day - 1 tablet every 8 hours.
  * Day 2: 500 mg of mefloquine, inside, in tablets of 250 mg 2 times a day - 1 tablet every 12 hours.
  * 3rd - 7th day: 250 mg of mefloquine, inside, in tablets of 250 mg 1 time a day at the same time.
  Interventions: Drug: Mefloquine
- group 1 cohort 2 (Experimental): 80 patients who receive Hydroxychloroquine prescribed according to the following scheme:
  • 1st day: 800 mg of hydroxychloroquine per day, inside, in 200 mg tablets, 2 tablets 2 times a day; 2nd - 7th day: 400 mg of hydroxychloroquine per day, inside, in tablets of 200 mg, 1 tablet 2 times a day.
  Interventions: Drug: Hydroxychloroquine
- group 2 cohort 1 (Experimental): A concomitant therapy consisting of Mefloquine in conjunction with azithromycin and tocilizumab will be given for 80 patients. Dosage of Mefloquine is same as for group 1 cohort 1.
  Interventions: Combination Product: Mefloquine + azithromycin + / - tocilizumab
- group 2 cohort 2 (Experimental): A concomitant therapy consisting of Hydroxychloroquine in conjunction with azithromycin and tocilizumab will be given for 80 patients. Dosage of Hydroxychloroquine is same as for group 1 cohort 2.
  Interventions: Combination Product: Hydroxychloroquine + azithromycin + / - tocilizumab

INTERVENTIONS:
Drug: Mefloquine — 1st day: 750 mg of mefloquine per day, inside, in tablets of 250 mg 3 times a day - 1 tablet every 8 hours.
  * Day 2: 500 mg of mefloquine, inside, in tablets of 250 mg 2 times a day - 1 tablet every 12 hours.
  * 3rd - 7th day: 250 mg of mefloquine, inside, in tablets of 250 mg 1 time a day at the same time.
  Arms: group 1 cohort 1
Drug: Hydroxychloroquine — 1. st day: 800 mg of hydroxychloroquine per day, inside, in 200 mg tablets, 2 tablets 2 times a day;
  2. nd - 7th day: 400 mg of hydroxychloroquine per day, inside, in tablets of 200 mg, 1 tablet 2 times a day.
  Arms: group 1 cohort 2
Combination Product: Mefloquine + azithromycin + / - tocilizumab — 1st day: 750 mg of mefloquine per day, inside, in tablets of 250 mg 3 times a day - 1 tablet every 8 hours.
  * Day 2: 500 mg of mefloquine, inside, in tablets of 250 mg 2 times a day - 1 tablet every 12 hours.
  * 3rd - 7th day: 250 mg of mefloquine, inside, in tablets of 250 mg 1 time a day at the same time.
  Arms: group 2 cohort 1
Combination Product: Hydroxychloroquine + azithromycin + / - tocilizumab — 1. st day: 800 mg of hydroxychloroquine per day, inside, in 200 mg tablets, 2 tablets 2 times a day;
  2. nd - 7th day: 400 mg of hydroxychloroquine per day, inside, in tablets of 200 mg, 1 tablet 2 times a day.
  Arms: group 2 cohort 2

SUMMARY:
Study of the effectiveness and safety of the drug Mefloquine, tablets 250 mg, produced by FSUE "SPC" Farmzaschita " FMBA of Russia (Russia), in comparison with the drug Hydroxychloroquine, tablets 200 mg, for the treatment of patients with coronavirus infection, in the "off-label" mode, to make a decision on the possibility of expanding the indications for use.

DETAILED DESCRIPTION:
Purpose of the study:

Study of the effectiveness and safety of the drug Mefloquine, tablets 250 mg, produced by FSUE "SPC" farmzaschita " FMBA of Russia (Russia), in comparison with the drug Hydroxychloroquine, tablets 200 mg, for the treatment of patients with coronavirus infection, in the "off-label" mode, to make a decision on the possibility of expanding the indications for use.

Study aims:

1. To study the efficacy of the drug Mefloquine, tablet 250 mg, for the treatment of patients with coronavirus infection (light and medium-heavy form), the appointment in the "off-label" in comparison with the drug Hydroxychloroquine tablets 200 mg, when administered in the mode "off label".
2. To study the effectiveness of the drug Mefloquine, tablet 250 mg, when administered in the mode "off label", in comparison with the drug Hydroxychloroquine tablets 200 mg, when administered in the mode "off label" when applied to a schema for the treatment of patients with severe coronavirus infection.
3. Evaluate the safety and tolerability of Mefloquine, 250 mg tablets, and Hydroxychloroquine, 200 mg tablets, for the treatment of patients with coronavirus infection (mild and moderate-severe forms).
4. Evaluate the safety and tolerability of Mefloquine, 250 mg tablets, and Hydroxychloroquine, 200 mg tablets, for the treatment of patients with coronavirus infection (severe forms), when used as part of a regimen for the treatment of patients with severe coronavirus infection.

Study design:

An open, randomized, multicenter comparative study of the efficacy and safety of Mefloquine and Hydroxychloroquine in "off-label" mode for the treatment of patients with COVID-19 coronavirus infection

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 years and older COVID19 positive confirmed by PCR, without ARDS and sepsis.
* Hospitalization of the patient.
* Signed informed consent for participation in the study.

Exclusion Criteria:

* The criteria for retiring a volunteer during the screening period are:

  1. Revoking informed consent of patients.
  2. Non-compliance of the volunteer with the inclusion criteria.
  3. First identified the condition and/or disease described in the criteria for inclusion.
  4. Positive test for HIV infection, Hepatitis B, C, syphilis.

The criteria for early termination of participation of volunteers in the study during the period of use of the study drug are:

1. Withdrawal of informed consent by a volunteer.
2. First identified the condition and/or disease described in the criteria for inclusion.
3. Occurrence of serious adverse events.
4. Adverse events that do not meet the criteria of severity, in the development of which, in the opinion of the researcher, further participation in the study may be harmful to the health or well-being of the volunteer.
5. The need for patients included in the study, antibiotics of the fluoroquinolone group.
6. Administrative reasons (termination of the study by the Sponsor or regulatory authorities), as well as gross violations of the Protocol that may affect the results of the study.
7. the Patient receives / needs additional treatment that may affect the outcome of the study or the patient's safety
8. Individual intolerance to research drugs
9. Erroneous inclusion (for example, the patient was included in violation of the criteria for inclusion/non-inclusion of the Protocol).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 320 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
1st primary endpoint for group 1 | up to 10 days
  The number of patients with development of respiratory failure requiring transfer to the ICU.
2nd primary endpoint for group 1 | up to 10 days
  The period of clinical recovery.
1st primary endpoint for group 2 | up to 10 days
  The period of clinical recovery.
2nd primary endpoint for group 2 | through study completion, an average of 3 months
  Frequency of fatal outcomes associated with coronavirus infection disease (COVID19)

SECONDARY OUTCOMES:
1st secondary endpoint for group 1 | on days 5 and 10
  A change in viral load by conducting PCR assay through different timeframes
2nd secondary endpoint for group 1 | on day 10
  Frequency of clinical cure on day 10 from the start of therapy
3d secondary endpoint for group 1 | up to 10 days
  The retention time of the reaction temperature from the start of the treatment.
4th secondary endpoint for group 1 | up to 10 days
  Concentration of C-reactive protein in blood plasma.
5th secondary endpoint for group 1 | up to 10 days
  Respiratory index.
6th secondary endpoint for group 1 | up to 10 days
  Frequency appearance unwanted phenomena and serious unwanted phenomena
1st secondary endpoint for group 2 | on days 5 and 10
  A change in viral load by conducting PCR assay through different timeframes
2nd secondary endpoint for group 2 | up to 10 days
  Respiratory index.
3d secondary endpoint for group 2 | up to 10 days
  The retention time of the reaction temperature from the start of treatment.
4th secondary endpoint for group 2 | up to 10 days
  Concentration of C-reactive protein in blood plasma.
5th secondary endpoint for group 2 | up to 10 days
  Number of patients required transition to alternative therapy schedule
6th secondary endpoint for group 2 | up to 10 days
  Frequency of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Astrelina, MD PhD,DSc., Principal Investigator — Burnasyan FMBC SRC FMBA of Russia
Locations (1):
- Burnasyan Federal Medical Biophysical Center FMBA of Russia, Moscow, Russia